CLINICAL TRIAL: NCT05948683
Title: Effects of Familiarity on Prosocial Effects of MDMA
Brief Title: Prosocial Effects of MDMA
Acronym: PEM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IRB23-0219; 5R01DA002812-35 (NIH)
Record Dates: First submitted 2023-06-30; First posted 2023-07-17 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2023-08

CONDITIONS: MDMA ('Ecstasy'); Social Interaction
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Familiar partner with placebo (Experimental): Participant engages in social interaction with 'familiar' partner under placebo
  Interventions: Drug: Placebo
- Familiar partner with MDMA (Experimental): Participant engages in social interaction with 'familiar' partner under MDMA
  Interventions: Drug: MDMA
- Unfamiliar partner with placebo (Experimental): Participant engages in social interaction with 'unfamiliar' partner under placebo
  Interventions: Drug: Placebo
- Unfamiliar partner with MDMA (Experimental): Participant engages in social interaction with 'unfamiliar' partner under MDMA
  Interventions: Drug: MDMA

INTERVENTIONS:
Drug: MDMA — The stimulant MDMA
  Arms: Familiar partner with MDMA; Unfamiliar partner with MDMA
Drug: Placebo — Dextrose
  Arms: Familiar partner with placebo; Unfamiliar partner with placebo

SUMMARY:
In this study, the aim is to test the hypothesis that MDMA produces greater prosocial effects when administered in the presence of a familiar, compared to an unfamiliar, person

DETAILED DESCRIPTION:
MDMA has shown promise as an adjunct to psychotherapy in the treatment of PTSD and other disorders. When used clinically with psychotherapy, the drug is believed to interact with the interpersonal components of the psychotherapy, especially the patient-therapist interaction. Indeed, patients and therapists usually form a strong alliance during several preparatory sessions, even before a drug is administered. Experts believe that the patient's familiarity and trust of the therapist is critical to the success of the intervention. Whereas therapeutic alliance is critical to the success of any psychotherapy, it may be especially important when psychoactive drugs are part of the treatment. The importance of this trust-building component preceding drug-assisted therapy has not been investigated.

There are mechanistic reasons to expect that MDMA will be more effective when a patient interacts with a familiar and trusted other person, compared to a stranger. MDMA is thought to exert its "prosocial" effects by increasing the social bonding hormone, oxytocin, and this hormone may contribute to its therapeutic effects. However, there is evidence that oxytocin increases feelings of connectedness specifically with familiar "in-group" members, and that it may not produce affiliative effects with individuals who are unfamiliar, or perceived to be outside their groups. Thus, the pro-social effects of oxytocin may depend on the degree of familiarity and closeness of the interacting partner. As noted above, during preparatory sessions in drug-assisted psychotherapy the patient forms a bond with a therapists before the drug is administered, which may serve to increase the 'in-group' effect of the drug, and thus maximize the therapeutic potential of the MDMA.

Controlled laboratory studies (without psychotherapy) show that MDMA produces prosocial effects on measures of mood and socio-emotional function. However, most of these studies are conducted in isolated individuals, or with study partners who have no prior relationship with the participant. In this proposed study the study team will investigate whether the prosocial effects of MDMA are greater when interacting with a partner to whom the participant feels close and more connected, compared to a partner who is unfamiliar.

To establish familiarity in one of the study groups the study team will use a procedure designed to establish feelings of closeness and connectedness between two strangers. In this procedure, two same-sex partners, who are initially strangers, engage in a 45 min conversation with one of two sets of topics provided by the experimenter. In one condition the topics remain superficial ("small talk" condition) and in the other, they become progressively deeper ("deep talk" condition) over the 45 mins. The study team and others have shown that the deep talk condition produces feelings of connection between the partners, and participants report feeling understood and liking their partners.

In the present study, the investigator will use this procedure to establish familiarity between conversation partners. The investigator aims to test the hypothesis that MDMA produces greater prosocial effects when administered in the presence of a familiar, compared to an unfamiliar, person. Participants will participate in four sessions, in which they receive MDMA (100 mg) or a placebo and then engage in a 15-min conversation with a familiar or unfamiliar person.

ELIGIBILITY:
Inclusion Criteria:

* used MDMA or psychedelic between 1-40
* high school diploma or equivalent
* BMI between 19 and 30
* verbal fluency in English

Exclusion Criteria:

* History of adverse effects with MDMA
* High blood pressure
* Any medical condition requiring regular medication
* Individuals with a current (within the last year) DSM-IV Axis 1 diagnosis
* Women who are pregnant or trying to become pregnant.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Natural Language Processing using large language model | during 15 minute test conversation, occurring 1.5 hours after drug administration
  Differences in speech content across all conditions
Facial expression analysis using HUMEAI software | during 15 minute test conversation, occurring 1.5 hours after drug administration
  Changes in emotional expressions during conversations

SECONDARY OUTCOMES:
Oxytocin | 120 minutes post drug administration
  Changes in oxytocin levels across all conditions
Self-reported feelings of connection using Likert scale conversation questionnaires | Collected at the end of the session, 240 minutes post-drug administration
  ratings of connectedness
Affective touch | Post-drug, 2 hours post-drug administration
  Ratings of pleasantness, intensity and want more touch (1-7) after differing velocities of touch

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided